CLINICAL TRIAL: NCT06718972
Title: Database of Real-world Study on the Treatment of Non-small Cell Lung Cancer With Leptomeningeal Metastasis in China
Brief Title: A Real-world Study on the Treatment of Non-small Cell Lung Cancer With Leptomeningeal Metastasis in China
Acronym: CLM-tree datab
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Haihong Yang, MD, Pricipal investigator, Chief Physician, Guangzhou Medical University
Other Study IDs: ES-2024-K125-02
Record Dates: First submitted 2024-11-27; First posted 2024-12-05 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Meningeal Metastasis; Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; meningeal metastasis; real-world study; database
MeSH Terms: conditions — Meningeal Carcinomatosis; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable- observational study — This is a retrospective and observational study. Not Applicable

SUMMARY:
This is a retrospective and prospective study planned to include NSCLC patients with Leptomeningeal metastasis (LM) and treated with antitumor therapy after 2018, from multiple centers such as the First Affiliated Hospital of Guangzhou Medical University, Guangdong Sanjiu Brain Hospital, etc., aiming to establish a database related to the treatment strategies of LM patients, and to evaluate the efficacy (eg. Overall Survival/Time to Failure) and safety of different treatment strategies of LM patients, etc., as well as the significance of concomitant testing in LM patients.

DETAILED DESCRIPTION:
retrospective and prospective study

ELIGIBILITY:
Inclusion Criteria:

* non-small cell lung cancer patients with Leptomeningeal metastases diagnosed after January 2018;
* Patients who underwent antitumor therapy after diagnosis of LM.

Exclusion Criteria:

* Patients with small cell lung cancer components;
* complicated with tumors other than non-small cell lung cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: non-small cell lung cancer patients with Leptomeningeal metastases
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | 6 years

SECONDARY OUTCOMES:
Time to failure(TTF) | 6 years
Change in cerebrospinal fluid and metabolic markers during treatment | 6 years
Safety during actual clinical treatment | 6 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Guangdong Sanjiu Brain Hospital, Guangzhou, Guangdong
  - the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong